CLINICAL TRIAL: NCT03180086
Title: Breast Cancer Risk Assessment in Women Aged 40-49
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Mara Schonberg, Principle Investigator - Staff Physician, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017P000129
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer risk; Primary Care; Women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer risk report (Experimental): An individualized report will inform women of their 5-year breast cancer risk using BCRAT or Tice (when breast density is available from a past mammogram), whichever is higher, and the average 5-year risk for women their age. The report will present 5-year risk as a frequency and in a pictograph and it will describe what experts recommend in terms of mammography screening, breast cancer prevention medications, breast MRIs, and BRCA testing, for women in their 40s based on their risk.
  Interventions: Other: Breast cancer risk report

INTERVENTIONS:
Other: Breast cancer risk report — An individualized report will inform women of their 5-year breast cancer risk using BCRAT or Tice (when breast density is available from a past mammogram), whichever is higher, and the average 5-year risk for women their age. The report will present 5-year risk as a frequency and in a pictograph and it will describe what experts recommend in terms of mammography screening, breast cancer prevention medications, breast MRIs, and BRCA testing, for women in their 40s based on their risk.

SUMMARY:
In a randomized controlled trial, the investigators will test the effect of a novel strategy for breast cancer risk assessment and risk-based management of women in their 40s seen in primary care. The investigators anticipate that this approach will lead to more optimal use of mammography screening and breast cancer prevention interventions in women in their 40s and as a result will improve care of these women.

DETAILED DESCRIPTION:
There is currently no standardized practice for addressing breast cancer risk in primary care. While there are guidelines encouraging PCPs to assess patients' breast cancer risk, few PCPs assess patients' risk due to time constraints in primary care, lack of familiarity with risk calculators, and knowledge on how to incorporate risk into the care of women. Around 20% of PCPs have reported using a risk calculator but few routinely asses patients' risk. In HealthCare Associates (HCA), Beth Israel Deaconess Medical Center's primary-care based practice, the online medical record (OMR) has recently been edited to allow for PCPs to enter patients' breast cancer risk. However, it is not known whether PCPs are using this tab. To calculate patient's breast cancer risk, PCPs must go to web-based calculators, ask patients their risk factors, enter the information and then add the estimated risk to OMR. Previous studies suggest that leaving risk assessment to PCPs results in few women having their risk assessed. Instead, PCPs tend to simply use family history when deciding whether or not patients are at high risk. However, family history is only one risk factor for breast cancer. Therefore, the investigators will send women ages 40-49 participating in this study a questionnaire to complete before a visit to assess their risk factors for breast cancer. Using this information, the investigators will calculate patients' breast cancer risk using the available breast cancer risk assessment models and will present women with a personalized breast cancer risk report immediately before a visit with their PCP. After the visit, patients will be asked to complete a follow-up questionnaire about their experience and through their medical records will be followed to learn whether or not they are screened with mammography. The investigators will follow high-risk women to learn whether or not they receive a screening breast MRI, BRCA gene testing, and/or the option to take breast cancer prevention medications. The investigators aim to recruit 445 women 40-49 years seen at HCA into a single arm trial to learn the effect of our personalized risk based approach to breast cancer screening and prevention on women in their 40's intentions to be screened and knowledge of the pros and cons of screening.

Specific Aims: To determine the effect of a personalized risk based approach for breast cancer screening and prevention for women in their 40s seen in primary care on:

1. women's intentions to be screened with mammography (primary outcome),
2. knowledge of the pros and cons of mammography screening, and
3. decisional conflict around screening; and on
4. patient report of PCP discussion of their breast cancer risk and of the pros and cons of mammography screening.

ELIGIBILITY:
Inclusion Criteria:

* women
* aged 40-49 years
* read and speak English
* scheduled for a routine visit or physical examination with a non-resident PCP in the next 4-12 weeks at HealthCare Associates (HCA, BIDMC's outpatient primary care practice).

Exclusion Criteria:

* women scheduled for acute care
* women who had or will have a mammogram within 6 months of their PCP visit
* women with a history of breast cancer or a BRCA mutation
* women already receiving screening breast MRIs
* women who have been referred to genetic counseling
* women who have taken or are taking tamoxifen or aromatase inhibitors for breast cancer prevention
* women with a history of an abnormal mammogram in the past two years
* women with a history of breast enlargement or reduction.

Ages: 40 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 338 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Screening intentions | 1 week
  Change in women's intentions to be screened with mammography after the intervention by 5-year breast cancer risk using a multivariable linear regression to examine the association between 5-year breast cancer risk and intentions to be screened after the intervention (as a continuous variable from 1 [not intending to be screened] to 15 [strongly intending to be screened]) adjusting for intentions to be screened at baseline as well as age, educational attainment, and race/ethnicity.

SECONDARY OUTCOMES:
Screening intentions within risk groups | 1 week
  The investigators will us the paired t-test (or Wilcoxon Signed Rank Test if data are not normal) to examine the differences in intentions to be screened with mammography after the intervention within each risk group.
Knowledge of the pros and cons of mammography screening | 1 week
  The investigators will use the paired t-test (or Wilcoxon Signed Rank Test when data are not normal) to examine the effect of the intervention on participants' knowledge of the benefits and risks of mammography screening (mean score on knowledge test)
Decisional conflict scale | 1 week
  The DCS is a validated 16 item scale to measure uncertainty around a decision, whether one feels informed, clear about their personal values, and supported in their decision-making (Cronbach's alpha=0.78 to 0.92); scores range 0-100 and lower scores indicate less conflict.
Difference in PCP discussion of breast cancer risk | 1 week
  The investigators will use McNemar's test to examine patient reports of PCP discussions of breast cancer risk [yes/no] before and after the intervention.
Difference in PCP discussion of pros/cons of mammography screening | 1 week
  The investigators will use McNemar's test to examine patient report of PCP discussion of the pros and cons of mammography screening [yes/no] before and after the intervention.
PCP discussion of breast cancer prevention medications | 1 week
  The investigators will use descriptive statistics to examine the proportion of women with >1.7% 5-year breast cancer risk that report discussing breast cancer prevention medications with their PCP.
PCP documentation of discussions of breast cancer medications | 1 week
  The investigators will use descriptive statistics to examine the proportion of women with >1.7% 5-year breast cancer whose PCPs document discussions about breast cancer prevention medications on the day of the visit.
Prescription of breast cancer prevention medications | 6 months
  The investigators will use descriptive statistics to report proportion of women with >1.7% 5-year breast cancer risk who were prescribed breast cancer prevention medications through review of medication lists
Time until breast screening MRI | 6 months
  The investigators will use the log-rank test to examine time until breast screening MRI among women with >20% lifetime breast cancer risk by lifetime breast cancer risk score as a continuous variable.
Referral to genetic counseling | 6 months
  The investigators will examine the proportion of women who meet NCCN criteria for genetic counseling for a BRCA mutation that are referred for genetic counseling
Attended genetic counseling | 6 months
  The investigators will examine the proportion of women who meet NCCN criteria for genetic counseling for a BRCA mutation that meet with a genetic counselor
Time until next mammogram after intervention | 21 months
  The investigators will examine the time until next mammogram after our intervention stratified by women's 5-year risk of breast cancer (based on the Breast Cancer Risk Assessment Tool [BCRAT]/Tice model [whichever is higher]) using the log-rank test.
Date of mammogram(s) after intervention | 21 months
  The investigators will document the date of mammogram performed on any women in the study during the study's follow-up time period.
Type of mammogram(s) after intervention | 21 months
  The investigators will document the type of mammogram performed on any women in the study during the study's follow-up time period.
No mammogram after intervention | 21 months
  The investigators will perform a chart review of women not identified as having had a mammogram during the study's follow-up time period to confirm that there is no mammogram noted in their screening sheet.
Risk report acceptability | 1 week
  The investigators will ask whether patients and PCPs found our risk report acceptable and/or helpful.
PCP facilitators and barriers | up to 24 months
  The investigators will examine facilitators and/or barriers noted by PCPs when assessing women's breast cancer risk and managing women based on their risk.
PCP risk of malpractice/litigation | up to 24 months
  The investigators will ask whether PCPs feel that our intervention would help lower their risk of malpractice litigation.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Schonberg, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schonberg MA, Davis RB, Karamourtopoulos MC, Pinheiro A, Sternberg SB, Jacobson AR, Aliberti GM, Mehta TS, Cluett JL, Cohen ML, Atlas T, Tung NM. A Pre-Test-Post-Test Trial of a Breast Cancer Risk Report for Women in Their 40s. Am J Prev Med. 2020 Sep;59(3):343-354. doi: 10.1016/j.amepre.2020.04.014. PMID 32828322